CLINICAL TRIAL: NCT07344181
Title: Efficacy of Liposomal Bupivacaine Scalp Nerve Block for Postoperative Pain Management After Supratentorial Craniotomy：a Randomized Controlled Trial
Brief Title: Efficacy of Liposomal Bupivacaine Scalp Nerve Block for Postoperative Pain Management After Supratentorial Craniotomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY2025-005-02
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Care
Keywords: Scalp nerve blocks，acute postoperative pain，Liposomal bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Preoperative scalp nerve block with liposomal bupivacaine.
  Interventions: Procedure: Preoperative scalp nerve block
- Control Group (Active Comparator): Preoperative scalp nerve block with 0.5% bupivacaine.
  Interventions: Procedure: Preoperative scalp nerve block

INTERVENTIONS:
Procedure: Preoperative scalp nerve block — Block of the supraorbital nerve, supratrochlear nerve, auriculotemporal nerve, zygomaticotemporal nerve, greater occipital nerve, and lesser occipital nerve.

SUMMARY:
This is a prospective, randomized, controlled trial conducted at Beijing Tiantan Hospital to evaluate the efficacy and safety of liposomal bupivacaine for scalp nerve block in managing postoperative pain after elective supratentorial craniotomy.

A total of 118 eligible patients (aged 18-64, ASA I-III) will be randomly assigned in a 1:1 ratio to one of two groups. The intervention group will receive a scalp nerve block using liposomal bupivacaine. The control group will receive a scalp nerve block using standard 0.5% bupivacaine. All patients will undergo standardized general anesthesia.

The primary outcome is postoperative pain intensity, measured by the Numerical Rating Scale (NRS) at multiple time points: 2, 12, 24, 48, and 72 hours after surgery. Secondary outcomes include the Glasgow Coma Scale (GCS) score, patient satisfaction, cumulative opioid consumption, and the incidence of adverse events.

The study aims to determine if a single administration of liposomal bupivacaine provides superior and prolonged analgesia compared to conventional bupivacaine, potentially improving pain management and recovery for craniotomy patients. The study duration is from October 2024 to May 2027.

DETAILED DESCRIPTION:
1. Background and Rationale:

   Postoperative pain following supratentorial craniotomy is a significant clinical concern, often requiring opioid-based analgesia. However, opioid use in neurosurgical patients is limited by side effects such as sedation, respiratory depression, and nausea, which can obscure neurological assessment and delay recovery. Scalp nerve blocks (SNBs) with local anesthetics like bupivacaine are a well-established component of multimodal analgesia for craniotomy, targeting the primary sources of postoperative pain-the pericranial muscles and scalp tissues. While effective, conventional bupivacaine provides analgesia for only up to 6-8 hours, leaving patients with inadequate pain control during the critical 72-hour postoperative period.

   Liposomal bupivacaine (LB) is an extended-release formulation designed to provide sustained analgesia for up to 72 hours. Its efficacy has been demonstrated in various surgical settings, but its application in neurosurgery, particularly for scalp nerve blocks, remains underexplored. This study aims to investigate whether a single preoperative scalp nerve block with liposomal bupivacaine can provide superior and prolonged analgesia compared to standard bupivacaine, thereby reducing opioid consumption and improving patient outcomes following craniotomy.
2. Objectives:

   Primary Objective: To compare the efficacy of liposomal bupivacaine versus standard bupivacaine for scalp nerve blocks in controlling postoperative pain, as measured by the Numerical Rating Scale (NRS) at 2, 12, 24, 48, and 72 hours after surgery.

   Secondary Objectives:

   To assess differences in cumulative opioid consumption postoperatively.

   To evaluate patient satisfaction using a standardized satisfaction scale.

   To monitor neurological status using the Glasgow Coma Scale (GCS).

   To record the incidence of adverse events (e.g., infection, hematoma, neurological deficits).
3. Study Design:

   Design: Prospective, single-center, randomized, controlled, parallel-group trial.

   Randomization: Eligible participants will be randomized in a 1:1 ratio to either the intervention group (liposomal bupivacaine) or the control group (standard 0.5% bupivacaine). Randomization will be performed using a computer-generated sequence.

   Blinding: Outcome assessors and data analysts will be blinded to group assignments. Due to the nature of the intervention, treating clinicians will not be blinded.
4. Participants:

   Inclusion Criteria:

   Adults aged 18-64 years.

   Scheduled for elective supratentorial craniotomy under general anesthesia.

   ASA physical status I-III.

   Preoperative GCS score of 15.

   Ability to provide informed consent.

   Exclusion Criteria:

   Chronic pain syndromes, opioid tolerance, or psychiatric disorders.

   Coagulopathy or infection at the block site.

   Allergy to local anesthetics.

   BMI <15 or >35.
5. Interventions:

   Intervention Group: Preoperative scalp nerve block with liposomal bupivacaine.

   Control Group: Preoperative scalp nerve block with 0.5% bupivacaine.

   Both groups will receive standardized general anesthesia and postoperative analgesia, including rescue opioids.
6. Outcome Measures:

   Primary Outcome: NRS pain scores at 2, 12, 24, 48, and 72 hours postoperatively.

   Secondary Outcomes:

   Opioid consumption (morphine equivalents).

   Patient satisfaction scores (5-point Likert scale).

   GCS scores.

   Adverse events related to the block or study drugs.
7. Sample Size:

   A total of 118 participants (59 per group) will be enrolled, accounting for a 20% dropout rate. This provides 90% power to detect a 25% difference in analgesia duration at a 5% significance level.
8. Statistical Analysis:

Data will be analyzed using SPSS v25.0. Continuous variables will be compared using t-tests or Mann-Whitney U tests; categorical variables will be analyzed with chi-square or Fisher's exact tests. Repeated-measures ANOVA will assess pain scores over time. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-64 years.

Scheduled for elective supratentorial craniotomy under general anesthesia.

ASA physical status I-III.

Preoperative GCS score of 15.

Ability to provide informed consent.

Exclusion Criteria:

* Chronic pain syndromes, opioid tolerance, or psychiatric disorders.

Coagulopathy or infection at the block site.

Allergy to local anesthetics.

BMI <15 or >35.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
NRS pain scores | 2, 12, 24, 48, and 72 hours postoperatively
  NRS pain scores at 2, 12, 24, 48, and 72 hours postoperatively.

SECONDARY OUTCOMES:
Opioid consumption | 2, 12, 24, 48, and 72 hours postoperatively.
  Opioid consumption (morphine equivalents)

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, Study Chair — Beijing Tiantan Hospital, Capital Medical University,Beijing, China
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this article will be shared following publication. The data will be available with researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Proposals should be directed to the corresponding author. Data requestors will need to sign a data access agreement to gain access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified IPD and supporting documents will become available starting 6 months after the publication of the primary trial results . The data will be accessible for a period of 5 years. This timeframe aligns with standard data sharing policies to ensure data are available while the research remains relevant.
Access Criteria: Who can access the IPD: Qualified researchers with a sound scientific proposal.
  What data will be accessible: De-identified individual participant data and the study protocol.
  How to access it: Proposals should be submitted to the corresponding author. Approved requestors will need to sign a data access agreement before gaining access via a secure file-sharing service.